CLINICAL TRIAL: NCT05670171
Title: Assessment the Safety and Efficacy of Debulking Atherectomy Versus Stent Angioplasty for Limb Ischaemia of Diabetic Lower Limb Atherosclerosis-occlusive Disease: A Multicenter, Randomized, Controlled Study.
Brief Title: Debulking Atherectomy Versus Stent Angioplasty for Limb Ischaemia of Diabetic Lower Limb Atherosclerosis-occlusive Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The Second Hospital of Hebei Medical University (Other); Shanxi Bethune Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); The Affiliated Hospital of Qingdao University (Other); Shanghai Pudong Hospital (Other); Tianjin Medical University General Hospital (Other); China-Japan Union Hospital, Jilin University (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DASALID
Record Dates: First submitted 2022-12-04; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Peripheral Arterial Disease
Keywords: Debulking Atherectomy; drug-coated balloon; Stent Angioplasty; Excimer laser atherectomy
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Debulking Atherectomy (Active Comparator): Excimer laser atherectomy combined with drug-coated balloon angioplasty
  Interventions: Procedure: Debulking Atherectomy
- Stent Angioplasty (Active Comparator): Nickel-titanium self-expanding bare stent
  Interventions: Procedure: Stent Angioplasty

INTERVENTIONS:
Procedure: Debulking Atherectomy — Excimer laser atherectomy combined with drug-coated balloon angioplasty
  Arms: Debulking Atherectomy
Procedure: Stent Angioplasty — Nickel-titanium self-expanding bare stent
  Arms: Stent Angioplasty

SUMMARY:
In order to assessment the safety and efficacy of debulking atherectomy versus stent angioplasty for limb ischaemia of diabetic lower limb atherosclerosis-occlusive disease, we intend to conduct a prospective, multicenter, randomized controlled, non-inferiority trial. The main surgical methods included stent angioplasty group (Nickel-titanium self-expanding bare stent) and debulking atherectomy group (Excimer laser atherectomy combined with drug-coated balloon angioplasty). The sample size was 244 patients, and the patients were followed up at 30 days, 180 days, and 365 days after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years old
2. Rutherford grade 2 to 5
3. Patients clinically diagnosed with arteriosclerosis obliterans of lower extremity (stenosis of lower extremity arteries greater than 70% or occlusion) and complicated with diabetes
4. The target vessel diameter ≥4mm
5. The total target length of the lesion is 30-210mm
6. The subject is able and willing to comply with all requirements, including 12-month follow-up and evaluation, voluntary participation and informed consen
7. Patients with ipsilateral iliac artery inflow tract patency (stenosis ≤50%) or ipsilateral iliac artery inflow tract lesions and successful management (residual stenosis < 30% after treatment, no severe (≥ grade D) flow-limiting dissection , no thrombosis, embolism or other serious adverse events)
8. Patients with at least one infrapopliteal artery for patency of the affected lateral foot before or after intraoperative treatment (stenosis ≤50%)

Exclusion Criteria:

1. Patients with vasculitis or Berger disease
2. Patients with contraindications to antiplatelet, anticoagulant and thrombolytic drugs
3. Patients who are allergic to contrast agents and nickel titanium materials
4. Patients with severe coagulation dysfunction or severe infection that is not under control and should not undergo surgery
5. Severe renal dysfunction (creatinine > 221umol/L)
6. Patients who received local or systemic thrombolytic therapy within 48 hours before surgery
7. Patients who had acute myocardial infarction within 30 days before surgery
8. Patients who had undergone major surgical procedures (heart, abdominal, or peripheral vascular open surgery) within 30 days before surgery
9. Patients who had a stroke within 6 months before surgery
10. Patients whose target arteries had received endovascular surgery within 14 days prior to surgery and patients who had other elective surgery plans during the study period
11. Patients with end-stage renal disease
12. Patients with previous major amputation of the target limb or restenosis after stent or bypass surgery for the target lesion
13. Patients with perforation, dissection, or other vascular injury requiring stenting or surgical operation in the approach or target vessel prior to enrollment
14. Patients with a life expectancy of < 12 months
15. A woman who is pregnant or breastfeeding
16. Patients who are participating in clinical trials of other drugs or devices that do not meet trial endpoints
17. Patients considered unsuitable for this trial by the investigators Exclusion criteria for angiography
18. Patients with severe calcification of the target lesions
19. Patients with aneurysms in the target vessels
20. Patients with acute or subacute thrombus in the target vessel
21. Patients with artificial vessels placed in the limb on the same side of the target vessel

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical-driven revascularization rate of target lesions 12-months after surgery | 12 months
  Clinically driven revascularization of target lesions was defined as a reduction of ABI ≥20% or >0.15 due to clinical symptoms or compared to the ABI after the initial surgery, any re-interventional therapy required for the target lesion.

SECONDARY OUTCOMES:
Technical success | Intraoperative
  Intraoperative angiography will demonstrated residual stenosis of the treated vessel <30%
Primary patency rate in patients with claudication (Rutherford grades 1-3) 12 -months after surgery | 12 months
  Primary patency was defined as peak systolic velocity ratio (PSVR) ≤2.4 (stenosis ≤50%) at 12-month follow-up.
The rate of unexpected major amputations 12 months after surgery in patients with severe ischemia (Rutherford grades 4-6) | 12 months
  The rate of unexpected major amputations 12 months after surgery in patients with severe ischemia (Rutherford grades 4-6)
Wagnar grade changes of diabetic foot ulcers at 6 months and 12 months after surgery (Rutherford Grade 4-6) | 6 months and 12 months
  Wagnar grade changes diabetic foot ulcers at 6 months and 12 months after surgery (Rutherford Grade 4-6)
Rutherford grades at 6 and 12 months postoperatively | 6 months and 12 months
  Rutherford grades at 6 and 12 months postoperatively
Changes in ankle-brachial index (ABI) at 6 and 12 months after surgery | 6 months and 12 months
  Changes in ankle-brachial index (ABI) at 6 and 12 months after surgery
The number of days of hospitalization | 1 month
  The number of days of hospitalization
The cost of hospitalization | 1 month
  The cost of hospitalization

OTHER OUTCOMES:
The incidence of surgery-related complications within 30 days after surgery | 30 days
  Including arterial dissection, perforation, rupture, embolism, acute thrombosis, pseudoaneurysm and hematoma formation.
All adverse events and serious adverse events were recorded during the study period. | 12 months
  All adverse events and serious adverse events were recorded during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Yongquan Gu, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (10):
- China (10):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - China-Japan Union Hospital, Jilin University, Changchun, Jilin
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Bethune hospital, Taiyuan, Shanxi
  - First Affiliated Hospital Xi'an Jiaotong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided